CLINICAL TRIAL: NCT06221462
Title: Neoadjuvant Sintilimab Plus Anlotinib Therapy in IB-IIIB Resectable Non-small Cell Lung Cancer (PRIORITY): a Prospective Single Center, Open Label, Phase II Study
Brief Title: Neoadjuvant Sintilimab Plus Anlotinib Therapy in IB-IIIB Resectable Non-small Cell Lung Cancer
Acronym: PRIORITY
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ningbo No.2 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBEY-HS-2023-008
Record Dates: First submitted 2023-12-26; First posted 2024-01-24 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non small cell lung cancer; Sintilimab; Anlotinib; neoadjuvant therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — sintilimab; anlotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment arm (Experimental)
  Interventions: Drug: Sintilimab; Drug: Anlotinib

INTERVENTIONS:
Drug: Sintilimab — 200mg, every 3 weeks, 3 cycles, in the neoadjuvant setting, and adjuvant 200mg,every 3 weeks no more than one year
Drug: Anlotinib — 8mg, orally, D1-14, every 3 weeks, 2 cycles in only neoadjuvant setting

SUMMARY:
This is a prospective single-center, open-label, phase II study evaluating the efficacy of sintilimab plus anlotinib as a neoadjuvant regimen in the treatment of IB-IIIB resectable non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Providing written informed consent prior to initiating the study.
2. Regardless of sex, aged ≥18 years and ≤75 years.
3. Histologically confirmed NSCLC.
4. At least one radiologically measureable lesion according to response evaluation criteria in solid tumors version 1.1(RECIST V1.1).
5. Treatment-naïve IB-IIIB resectable NSCLC (American Joint Committee on Cancer 8th tumor-node-metastasis classification).
6. Epidermal growth factor receptor(EFGR)/anaplastic lymphoma kinase(ALK)/ROS proto-oncogene 1(ROS1) wild type NSCLC.
7. Absence of bleeding risk.
8. Consent to surgical treatment.
9. Indication for surgery confirmed by surgeons.
10. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
11. Expected survival time more than 6 months.
12. Sufficient organ reserve, detailed as follows:(1) the absolute neutrophil count ≥1.5×109/L without the use of granulocyte colony-stimulating factor for the past 14 days prior to the first dose of study drugs;(2) platelet count ≥100×109/L without blood transfusion within the 2 weeks before the enrollment;(3) hemoglobin >9g/dL without recent usage of blood transfusion 14 days prior to the study;(4) total bilirubin ≤ 1.5 fold the upper limit of normal (ULN), or total bilirubin >1.5 fold ULN but direct bilirubin ≤ 1 fold ULN;(5) aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5×ULN;(6) blood creatinine ≤ 1.5 fold ULN and creatinine clearance (calculated by the Cockcroft-Gault formula) ≥ 60ml/min;(7) adequate coagulation function, defined by international normalized ratio (INR) or prothrombin time(PT) less than 1.5 fold ULN;(8) normal thyroid function defined by the normal range of thyroid-stimulating hormone (TSH); otherwise, abnormal level of TSH with normal range of T3(or Ft3) and Ft4;(8) cardiac enzyme profile within the normal limits (merely laboratory abnormity without clinical significance based on investigator's decision is allowed)
13. For female participants of childbearing age, a urine or serum pregnancy test should be performed within 3 days before receiving the first dose of the study drugs, and the result must be negative. If the urine pregnancy test result is inconclusive, a blood pregnancy test is warranted. Postmenopausal women are defined as those who have been without menstruation for at least 1 year, or have undergone surgical sterilization or hysterectomy.
14. In the presence of pregnancy risk, all participants (both male and female) are required to use contraceptive measures with an annual failure rate of less than 1% throughout the entire treatment period up to 120 days following the last dose of the study drugs.

Exclusion Criteria:

Exclusion criteria as follows：

1. Other malignancy rather than NSCLC diagnosed within 5 years prior to the first dose of the study given, except for definitively treated basal cell carcinoma, squamous cell carcinoma of the skin, and/or in situ carcinoma.
2. Enrolled in an ongoing interventional clinical trial, or receiving other study drugs or study medical devices within 4 weeks prior to the first dose of this study drugs.
3. A history of receiving the following therapies: anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death ligand-1 (anti-PD-L1) or anti-programmed cell death ligand-2 (anti-PD-L2) drugs, or drugs targeting T cell receptor (such as cytotoxic T-lymphocyte-associated protein 4, tumor necrosis factor receptor superfamily member 4 and CD137).
4. A history of receiving targeted therapy such as anti-vascular endothelial growth receptor (VEGR)/ vascular endothelial growth factor receptor (VEGFR), rapidly accelerated fibrosarcoma(RAF), mitogen-activated protein kinase(MAPK), platelet-derived growth factor Receptor(PDGFR) or fibroblast growth factor receptor(FGFR).
5. Receiving traditional Chinese medication or immunomodulatory drugs (including thymopentin, interferon, interleukin, except for controlling pleural effusion) as systemic therapy within 2 weeks prior to the first dose of the study drugs.
6. Active systemic auto-immune disease requiring systemic treatment within 2 years prior to the first dose of the study drugs, such as the use of disease-modifying drugs, glucocorticoids or immunosuppressants. Alternative therapies (such as thyroid hormone, insulin, or physiological glucocorticoids used for adrenal or pituitary insufficiency) are not considered as systemic treatment.
7. Systemic glucocorticoid therapy (excluding nasal, inhaled or other local routes of glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drugs.
8. Undergoing allogeneic organ transplant (excluding corneal transplantation) or allogeneic hematopoietic stem cell transplant.
9. Allergy to the active ingredient or excipients of the study drug, sintilimab.
10. Having not recovered from any toxicities and/or complications caused by prior interventions before the initiation of the study (i.e., ≤ Grade 1 or to baseline, excluding fatigue or hair loss)
11. Known history of human immunodeficiency virus (HIV) infection.
12. Untreated active hepatitis B (defined as hepatitis B surface antigen positive with detectable hepatitis B virus(HBV)-DNA copies exceeding the upper limit of normal values).
13. Active hepatitis C infection.
14. Receiving a live vaccine within 30 days prior to the first dose of the study drug.
15. Pregnant or lactating women.
16. Other investigator's defined uncontrolled systemic disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
major pathological response (MPR) | 10 days postoperatively
  Viable tumor cells are no more than 10% in the resected specimen

SECONDARY OUTCOMES:
pathological complete response (pCR) | 10 days postoperatively
  Viable tumor cells are not found in the resected specimen
treatment-related adverse events (TRAEs) | 90 days after the last dose of study drugs
  TRAEs including immune-related adverse reaction are documented and graded based on the US National Cancer Institute's Common Terminology Criteria for Adverse Events 5.0 criteria.
disease-free survival (DFS) | 5 years
  DFS is defined as the duration between the date of surgery and the date on which tumor recurrence is confirmed
rate of operative complications | 30 days postoperatively
  The rate of surgical complications (such as bleeding, bronchopleural fistula,ect) are recorded and graded according to Clavien-Dindo criteria
overall survival(OS) | 5 years
  OS is defined as the duration between the date of surgery and the date of all-cause death

OTHER OUTCOMES:
minimal residual disease (MRD) | 5 years
  MRD is evaluated by testing circulating tumor DNA (ctDNA) in peripheral blood sample using next-generation sequencing(NGS) method. Each participant will undergo a minium of 3 tests for MRD.

CONTACTS AND LOCATIONS:
Overall Officials: Guofang Zhao, MD, Principal Investigator — Ningbo No.2 Hospital

IPD SHARING:
Plan to Share IPD: No